CLINICAL TRIAL: NCT01955018
Title: Comparison of the Ultra-low-dose Veo Algorithm With the Gold Standard Filtered Back Projection for Detecting Pulmonary Asbestos-related Conditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHU-0166; 2012-A00618-35
Record Dates: First submitted 2013-09-02; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Asbestos-exposed Workers
Keywords: computed tomography; radiation; screening; asbestos; workers; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- VeoTM (Experimental): A new algorithm called VeoTM (General Electric Healthcare, Milwaukee, MI, USA) decreases the image noise up to 70% compared with the gold standard FBP model. Moreover, Veo improves spatial resolution with excellent detection of low and high contrast objects from a CT Dose Index (CTDIvol) equal to 0.3 mGy
  Interventions: Device: New algorithm called VeoTM (General Electric Healthcare, Milwaukee, MI, USA)
- gold standard FBP model (Other): The objective of the present study is to compare Veo with the gold standard FBP for detecting pulmonary asbestos-related conditions among workers previously exposed to asbestos. Comparisons included radiation delivered and image quality
  Interventions: Device: New algorithm called VeoTM (General Electric Healthcare, Milwaukee, MI, USA)

INTERVENTIONS:
Device: New algorithm called VeoTM (General Electric Healthcare, Milwaukee, MI, USA) — The objective of the present study is to compare Veo with the gold standard FBP for detecting pulmonary asbestos-related conditions among workers previously exposed to asbestos. Comparisons included radiation delivered and image quality.

SUMMARY:
Asbestos fibers were intensively used throughout the 20th century and remain prevalent in developing countries. However, asbestos exposure induces a variety of benign and malignant pleural and lung diseases. The most common asbestos-induced neoplasm is lung cancer. Moreover, thin-section computed tomography (CT) is more sensitive than a chest x-ray for detecting early asbestos-related conditions. Increased exposure to radiation underpins the consequences of cancer induction. However, reducing CT doses increases image noise from the filtered back projection (FBP) reconstruction. Strategies to reduce radiation exposure include the use of iterative reconstruction algorithms. A new algorithm called VeoTM (General Electric Healthcare, Milwaukee, MI, USA) decreases the image noise up to 70% compared with the gold standard FBP model. Moreover, Veo improves spatial resolution with excellent detection of low and high contrast objects from a CT Dose Index (CTDIvol) equal to 0.3 mGy.

The objective of the present study is to compare Veo with the gold standard FBP for detecting pulmonary asbestos-related conditions among workers previously exposed to asbestos. Comparisons included radiation delivered and image quality.

DETAILED DESCRIPTION:
Asbestos-exposed workers will be recruited following referral to our radiology department for the evaluation of asbestos-related disease. CT examinations will be performed with a 64-slice CT system (Discovery CT 750HD; GE Healthcare, Milwaukee, WI) and will consist of two successive acquisitions. Each examination, the normal-dose (FBP acquisition) and ultra-low-dose (Veo acquisition) spiral CT, will be performed in supine position, on the entire thorax, at full inspiration and without contrast agent injection.

In order to perform the two acquisitions without increasing radiation, standard acquisition will be performed with the same kV with mA equal to patient's body weight minus 10. To conserve image quality, 60 mA will be the inferior limit. The other CT parameters will be rotation time 0.5 s and pitch 1.375. Image data will be reconstructed with FBP algorithm.

The Veo acquisition will be performed with constant CT parameters including: a tube voltage of 100 kV, a tube current of 20 mA, pitch of 0.984 and rotation time 0.4 s. Image data will be reconstructed with the Veo algorithm.

Each CT acquisition will be viewed independently by two experienced radiologists (2 to 7 years of experience). The low-dose images with Veo reconstruction will be interpreted before the standard CT and on separate weeks to minimize recall bias. Then, the more experienced radiologist will evaluate the detection and characterization of pleuroparenchymal abnormalities by a second and simultaneous reading of the Veo and FBP acquisitions. Because FBP images are benchmark practice, when a lesion will be found only on Veo images, it will be regarded as a false positive.

The following asbestos-related pleural and parenchymal abnormalities will be recorded as present or absent. Pleural abnormalities considered will be: pleural plaques, diffuse pleural thickening and pleural effusion.

CT features of asbestosis will include subpleural dots and branching opacities, curvilinear subpleural lines, areas of ground glass opacities, septal lines, reticulations and honeycombing.

Presence of nodules will also be recorded. We will note for each abnormality: localization (side, table position) and nature (non-solid, part-solid, solid or calcified).

ELIGIBILITY:
Inclusion Criteria:

* asbestos-exposed workers
* ability to give a written informed consent

Exclusion Criteria:

* - previous history of cancer
* previous history of thoracic surgery
* other interstitial pathology known

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Pleural and parenchymal abnormalities | at day 1
  The kappa coefficient will be used to measure agreement for categorical parameters and Pearson's correlation coefficient and Lin concordance correlation coefficient for quantitative data.

SECONDARY OUTCOMES:
Radiation dose | at day 1
  The dose length product (DLP) will be recorded.
Quality images assessment | at day 1
  Respiratory artifacts will be graded on a three-point scale (1 = negligible, 2 = moderate, 3 = salient).
  Images noise will be studied in the axial and coronal planes. A similar scale will be used for subjective image quality in the mediastinum and parenchyma windows.
  Objective image noise (Standard Deviation) and average CT numbers (in Hounsfield's units) will be measured with circular regions of interest (ROI) on different anatomical levels, 10 mm in diameter.
  The signal to noise ratio (SNR) will also be calculated using the equation SNR = CT numbers / noise.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Tekath M, Dutheil F, Bellini R, Roche A, Pereira B, Naughton G, Chamoux A, Michel JL. Comparison of the ultra-low-dose Veo algorithm with the gold standard filtered back projection for detecting pulmonary asbestos-related conditions: a clinical observational study. BMJ Open. 2014 May 30;4(5):e004980. doi: 10.1136/bmjopen-2014-004980. PMID 24879827